CLINICAL TRIAL: NCT04403425
Title: Correlation of Central and Peripheral Measures of Tissue Perfusion During Emergency Laparotomy - a Pilot Study
Brief Title: Tissue Perfusion During Emergency Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mirjana Cihoric, MD, Research fellow, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-19069841
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Emergency Laparotomy; Intestinal Obstruction; Perforated Viscus
Keywords: emergency laparotomy; tissue perfusion; hemodynamic instability
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency laparotomy, obstruction: Patients undergoing emergency laparotomy for intestinal obstruction in need of intraoperative Noradrenaline infusion to maintain predefined normotension.
- Emergency laparotomy, perforation: Patients undergoing emergency laparotomy for perforated ventricle or intestine in need of intraoperative Noradrenaline infusion to maintain predefined normotension.

SUMMARY:
This study is investigating the effect of intraoperative Noradrenaline on cardiac preload and stroke volume, after initial fluid resuscitation, in order to assess whether there is a masked preload responsiveness and ultimately whether the correction of this potential preload-responsiveness with fluid therapy will translate into increased tissue perfusion in emergency laparotomy.

DETAILED DESCRIPTION:
Early detection and treatment of insufficient tissue perfusion and oxygenation is the main purpose of perioperative haemodynamic monitoring and management. Hypovolemia, septicaemia, and low flow states affecting central and peripheral perfusion are frequent in patients undergoing emergency laparotomy.

This study aims to assess the effects of Noradrenaline (NA) on cardiac preload, and tissue perfusion in patients undergoing emergency laparotomy, to investigate potential macro/microcirculatory uncoupling.

A single-centre, prospective interventional non-blinded single-arm study at the Department of Anaesthesiology and Intensive care Unit, Copenhagen University Hospital Hvidovre, Denmark. We will include patients undergoing emergency laparotomy. The study start is January 2021. After informed consent, patients will be included if they have an intraoperative need for Noradrenaline infusion >0.1 mcg/kg/min to maintain MAP ≥65 mmHg after resuscitation with a goal-directed fluid therapy algorithm. 20 patients will be included.

Intervention: At a steady state (MAP ≥65 mmHg) during the surgical procedure, we will reduce NA to investigate whether patients will be preload responsive while maintaining MAP > 50 mmHg and limiting stroke volume reduction to no more than 30%. After a subsequent fluid challenge, we will increase the dose of NA to re-establish a MAP ≥65 mmHg. In addition, peripheral and central perfusion indices, including gut perfusion, will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or over) undergoing emergency laparotomy/laparoscopy for following abdominal pathology:

   1. Perforated viscus
   2. Intestinal obstruction
2. Emergency re-operations after elective surgery owing to paralytic/obstructive ileus, anastomotic leakage
3. Provided verbal and written informed consent
4. Must speak and understand the Danish language
5. Intraoperative indication for Norepinephrine infusion

Exclusion Criteria:

1. Appendectomies, cholecystectomies, negative diagnostic laparoscopies/laparotomies, herniotomies without bowel resections, sub-acute internal hernias after gastric bypass surgery, sub-acute surgery for inflammatory bowel diseases.
2. Reoperation owing to fascial separation with no other abdominal pathology identified and sub-acute colorectal cancer-surgery will be excluded from the cohort. Sub-acute surgery is defined as surgery planned within 48 hours.
3. Intestinal Ischemia
4. intraabdominal bleeding
5. Traumas, gynecological, urogenital and other vascular pathology, pregnant patients.
6. Dementia and/or cognitive dysfunction (diagnosed). If the patient is not awake, alert, and oriented, times three (to person, place, and time), this also qualifies as an exclusion criterion.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include patients undergoing emergency laparotomy on suspicion of abdominal pathology, in need of intraoperative Noradrenaline infusion to maintain predefined normotension.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Preload dependency | intraoperatively (during general anesthesia)
  the incidence of preload dependency defined as stroke volume increase of >10% during fluid challenge after reduction of Noradrenaline.

SECONDARY OUTCOMES:
Tissue perfusion and fluid status | intraoperatively (during general anesthesia)
  changes in perfusion indices (delta values) after NA reduction, one fluid bolus, and subsequent restoration of blood pressure with Noradrenaline.
Tissue perfusion | intraoperatively (during general anesthesia)
  Other endpoints of interest are the correlation between gut perfusion and indices of central and peripheral perfusion (urethral, cerebral, tissue).

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No